CLINICAL TRIAL: NCT03353402
Title: Altering the Gut Microbiota of Melanoma Patients Who Failed Immunotherapy Using Fecal Microbiota Transplantation (FMT) From Responding Patients
Brief Title: Fecal Microbiota Transplantation (FMT) in Metastatic Melanoma Patients Who Failed Immunotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Gal Markel, Chief Scientist of The Ella Lemelbaum Institute of Immuno-Oncology, Principal Investigator, Associate Professor of Immunology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-17-3956-GM-CTIL
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Melanoma Stage Iv; Unresectable Stage III Melanoma
Keywords: Melanoma; Fecal Microbiota Transplantation; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplant (FMT) (Experimental): FMT includes a colonoscopy conducted by a gastroenterologist followed by stool capsules which will be swallowed by the patient.
  Interventions: Procedure: Fecal Microbiota Transplant (FMT)

INTERVENTIONS:
Procedure: Fecal Microbiota Transplant (FMT) — Patients with metastatic melanoma who responded to immunotherapy will serve as the fecal implant donors. The tested fecal implant will be used for two different products. The first part of the tested stool will be mixed with a saline solution, strained and infused into your bowel using colonoscopy. The second part of the tested stool will be packed into capsules. These stool capsules are at the size of standard drug-containing capsules and can be swallowed in a standard manner. Stool capsules are a common method of FMT and has been used worldwide for several years. After the colonoscopy, you will be asked to swallow the capsules. Swallowing the capsules will be conducted at the clinic, and does not require any additional procedures.

SUMMARY:
Altering the Gut Microbiota of Melanoma Patients Who Failed Immunotherapy Using Fecal Microbiota Transplantation (FMT) From Responding Patients.

FMT includes both colonoscopy and stool capsules.

DETAILED DESCRIPTION:
This is a phase I single-center study of fecal microbiota transplant (FMT) in melanoma patients who failed at least one line of PD-1 blockade.

Eligible patients must have a disease amenable to biopsy and lack of contra-indications to FMT.

Patients will undergo a baseline evaluation including imaging, tumor biopsy, blood samples and stool studies to confirm suitability for the study.

Eligible patients will undergo FMT. The FMT includes a colonoscopy followed by stool capsules.

Patients will undergo repeated evaluations including follow-up blood, stool and radiological testings.

The study will be conducted over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed diagnosis of metastatic melanoma.
* Failed at least one line of PD-1 blockade.
* ECOG Performance Status 0-2
* Able to provide written informed consent.

Exclusion Criteria:

* Presence of absolute contra-indications to FMT administration.
* Severe dietary allergies (e.g. shellfish, nuts, seafood).
* Anatomic contra-indications to colonoscopy.
* Inability to swallow capsules.
* Current participation in a study of an investigational agent.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy prior to trial treatment.
* History of bleeding disorder, chronic kidney disease, Inflammatory bowel disease.
* History of a major abdominal surgery
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of FMT-related Adverse Events | 4 years
  Number of patients with adverse events that emerged post FMT
Proper implant engraftment | 4 years
  Comparing of the patients' gut bacterial composition pre and post-FMT and in relation to their donors. Bacterial composition will be quantified by the operational taxonomic unit (OTU) in the stool

SECONDARY OUTCOMES:
Changes in composition of immune cell population | 4 years
  Changes in the relative abundance of different immune cell population (such as the proportion of CD8+ T cells) pre and post-FMT.
Changes in activity of immune cells | 4 years
  Changes in levels of proteins that represent immune activity against cancer (such as measurements of blood interferon gamma levels), pre and post FMT

OTHER OUTCOMES:
Objective Response Rate (ORR) | 4 years
  Number of patients with objective responses divided by the total number of evaluable patients, according to imaging studies (RECIST 1.1) and iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Markel, MD, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Villemin C, Six A, Neville BA, Lawley TD, Robinson MJ, Bakdash G. The heightened importance of the microbiome in cancer immunotherapy. Trends Immunol. 2023 Jan;44(1):44-59. doi: 10.1016/j.it.2022.11.002. Epub 2022 Dec 1. PMID 36464584